CLINICAL TRIAL: NCT04222725
Title: A Multicenter, Double-Masked, Randomized, Vehicle-controlled, Dose-ranging Study to Evaluate the Safety of TRS01 Eye Drops in Participants With Post-surgical Inflammation
Brief Title: A Study of TRS01 in Participants With Post-surgical Ocular Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tarsier Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tarsius 2020; 2019-004327-20 (EudraCT Number); Grant Agreement Number 879598 (Other Grant/Funding Number: European Union's Horizon 2020)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-01

CONDITIONS: Post Surgical Ocular Inflammation
Keywords: postoperative; postsurgical; ocular; inflammation; pain
MeSH Terms: conditions — Inflammation; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TRS01 low dose (Experimental)
  Interventions: Drug: TRS01 eye drops
- TRS01 medium dose (Experimental)
  Interventions: Drug: TRS01 eye drops
- TRS01 high dose (Experimental)
  Interventions: Drug: TRS01 eye drops
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo eye drops

INTERVENTIONS:
Drug: TRS01 eye drops — Dosed 4 times a day (QID)
  Arms: TRS01 low dose
Drug: TRS01 eye drops — Dosed QID
  Arms: TRS01 medium dose
Drug: TRS01 eye drops — Dosed QID
  Arms: TRS01 high dose
Drug: Placebo eye drops — Dosed QID
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and preliminary efficacy of TRS01 eye drops as compared to placebo on participants with ocular inflammation after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Pre-operatively, individuals of either gender or any race will be eligible for study participation if they are:

* 18 years of age or older.
* Able to provide informed consent, follow instructions and complete all required study visits for the duration of the study.
* Scheduled for routine cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens (IOL) implantation, and not combined with any other surgery.
* Have vision ≥ 20/200 in the non-study eye.
* Able to self-administer eye drops (tested during screening by self-administration of "artificial tears"), or have a care provider that can administer the drops.
* Have no known sensitivity /allergy to the TRS01 or formulation excipients.
* Using adequate birth control by men and women, if of reproductive potential and sexually active, as specified per protocol
* Randomization inclusion criteria as specified per protocol.

Exclusion Criteria:

* Scheduled to undergo cataract surgery in the non-study eye for the duration of the study.
* Receiving specific medication/interventions as specified per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Inglewood, Inglewood, California
  - Petaluma, Petaluma, California
  - Washington, MO, Washington, Missouri
  - New York, New York, New York
  - Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRS01 Low Dose | TRS01 Medium Dose | TRS01 High Dose | Placebo
Started | 8 | 10 | 9 | 10
Completed | 8 | 9 | 9 | 10
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRS01 Low Dose | TRS01 Medium Dose | TRS01 High Dose | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 9 | 10 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 0 | 4 | 13
  >=65 years | 4 | 5 | 9 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.11) | 63.8 (7.77) | 74.9 (5.84) | 67.0 (7.79) | 67.6 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 7 | 26
  Male | 2 | 3 | 3 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 5 | 7 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Dark Brown | 5 | 5 | 5 | 8 | 23
  Light Brown | 0 | 1 | 2 | 0 | 3
  Blue | 3 | 2 | 2 | 1 | 8
  Gray | 0 | 1 | 0 | 0 | 1
  Hazel | 0 | 1 | 0 | 1 | 2
Anterior Chamber Cell Grade in the Study Eye [Count of Participants; unit: Participants] — The following scoring scale for anterior chamber cells was used:
  0 = No cells seen
  1. = 1 - 5 cells
  2. = 6 - 15 cells
  3. = 16 - 30 cells
  4. = greater than 30 cells There is a direct correlation between the number of cells and severity of the disease
  Participants
    2 (6-15 Cells) | 3 | 3 | 3 | 4 | 13
    3 (16-30 Cells) | 3 | 6 | 3 | 4 | 16
    4 (>30 Cells) | 2 | 1 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Both Systemic and Ocular Adverse Events
Description: Number of adverse events that occurred during the study
Time Frame: 14 days
Population: All randomized subjects who took at least 1 dose of study drug
Measure: Number; unit: Number of TEAE
Arm/Group | TRS01 Low Dose | TRS01 Medium Dose | TRS01 High Dose | Placebo
Number analyzed (Participants) | 8 | 10 | 9 | 10
Number of TEAE | 0 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Safety Population: all randomized subjects who took at least 1 dose of study drug. Adverse events were collected from the signing of the Informed Consent Form (Screening) to the end of study (Day 15 or Early Termination).
Arm/Group | TRS01 Low Dose | TRS01 Medium Dose | TRS01 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 2/10 | 0/9 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRS01 Low Dose (N=8) | TRS01 Medium Dose (N=10) | TRS01 High Dose (N=9) | Placebo (N=10)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Device Dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Principal Investigators (and their Institutions) and the Sponsor that restricts the PI's rights to discuss or publish results of this study without the prior written consent of the study Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04222725/Prot_SAP_000.pdf